CLINICAL TRIAL: NCT06294717
Title: The Effect of Progressive Relaxation Exercises on Physiological Parameters, Pain and Anxiety After Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Neslihan Atli, Midwife, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkUPhStudentNeslihanATLI
Record Dates: First submitted 2024-02-24; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Progressive relaxation exercises will be explained and taught to the puerperant after cesarean section. Experimental Group (in the group where progressive relaxation exercises were applied); The first application will be made at the 8th postoperative hour. Before the application, the Puerperal Identification Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled out. Starting from the 8th post-op hour, the first, second and third applications will be made eight hours apart within a 48-hour period. On the second day, progressive relaxation exercises will be performed once, twice and three times at eight-hour intervals. At the end of the second day, the Postpartum Definition Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled in again.
  Interventions: Other: Progressive relaxation exercises will be applied.
- Control Group (No Intervention): No application will be made with participants in the control group. At the 8th postoperative hour, the Puerperal Identification Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled out. These participants will be asked not to engage in regular physical activity or sports for 2 days and not to make any changes in their living habits.
  During the interview two days later, the Postpartum Identification Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled out again by the postpartum women.

INTERVENTIONS:
Other: Progressive relaxation exercises will be applied. — Progressive relaxation exercises will be not applied.
  Arms: Experimental Group

SUMMARY:
Caesarean section is a surgical procedure that can be performed before or during birth in cases where the life of the mother and fetus is threatened or upon the request of the mother and father. One of the most common problems after cesarean section is abdominal pain. Progressive relaxation exercises are a method that allows certain muscle groups in the body to first contract and then relax. Progressive relaxation exercises have been proven to have positive effects on anxiety. By applying progressive relaxation exercises, the parasympathetic nervous system is activated; Thus, heart and respiratory rate and blood pressure can be kept within normal limits. This study will be conducted to determine the physiological parameters, pain and anxiety levels of progressive relaxation exercises, one of the non-pharmacological methods, on women giving birth by cesarean section.

DETAILED DESCRIPTION:
Purpose of the research: (Must be clearly stated and compatible with the subject title) It will be carried out as a randomized controlled experimental design to determine the effect of progressive relaxation exercises on physiological parameters, pain and anxiety after cesarean section.

10. Materials and methods of the research: Type of Study: This research is a randomized controlled study.

Research Questions/Hypotheses:

Hypothesis 1 (H1): Progressive relaxation exercises after cesarean section have an effect on physiological parameters.

Hypothesis 2 (H1): Progressive relaxation exercises after cesarean section have no effect on physiological parameters.

Hypothesis 3 (H2): Progressive relaxation exercises have an effect on pain after cesarean section.

Hypothesis 4 (H2): Progressive relaxation exercises have no effect on pain after cesarean section.

Hypothesis 5 (H3): Progressive relaxation exercises after cesarean section have an effect on anxiety.

Hypothesis 6 (H3): Progressive relaxation exercises have no effect on anxiety after cesarean section.

Location and Characteristics of the Research: The research will be conducted between September 1, 2023 and August 1, 2024, in the gynecology service of Şanlıurfa Training and Research Hospital, with women who gave birth by cesarean section and meet the inclusion criteria. This hospital was chosen due to its nature as a regional hospital and the density of cesarean births.

Population-sample of the research: The population of this research will consist of women who gave birth by cesarean section in the gynecology service of Şanlıurfa Training and Research Hospital between February 1, 2024 and August 1, 2024, 2024. Taking into account the tests to be used to calculate the minimum sample size to be included in the study, GPower analysis was performed and the sample size was calculated as 120 puerperal mothers. A total of 120 postpartum women will be included in the sampling, including 60 postpartum women who meet the inclusion criteria for the study, who agree to participate in the study, and who gave birth by cesarean section to which progressive relaxation exercises are applied, and 60 postpartum women who give birth by cesarean section to which progressive relaxation exercises are not applied.

Data Collection Forms and Tools:

Postpartum Identification Form:

This form was prepared and developed by the researchers based on the literature. It consists of questions to determine sociodemographic, medical and obstetric characteristics.

Beck Anxiety Scale: Developed by Beck et al. in 1988, the scale measures the frequency of anxiety symptoms experienced by a person. The person is asked to indicate how much the listed anxiety symptoms bother him or her in the last week. The scale, consisting of twenty-one items, provides a four-point Likert type measurement (0 being not at all, 3 being seriously). It was used in the study to evaluate the overlap validity of typical anxiety symptoms. Turkish validity and reliability study was conducted by Ulusoy, Şahin and Erkmen in 1998. The scale consists of items containing somatic symptoms and subjective anxiety. (Cronba alpha value=0.93)

Visual Analog Scale (VAS):

It is a pain level measurement method created by Albersnagel (1988). It is used to make the undetermined feeling of pain numerically meaningful. The validity and reliability study in our country was conducted by Aydin et al. (2011). The range of 0 (zero) and 10 cm is determined on a ruler. 0 (zero) means "no pain" and 10 means "worst possible pain". The patient is asked to mark the place that expresses his pain on the line. The distance marked by the patient is measured by taking the zero starting distance. The benefit of the Visual Comparison Scale is that it is a proven scale and has been shown to be sensitive to changes in a patient's pain experience. It is quick to use and relatively easy to understand for most patients. It avoids the misuse of descriptive words to describe pain and allows meaningful comparison of measurements over time.

Physiological Parameters:

Physiological Measurements Form; vital signs of the woman giving birth; It is a chart where pulse, respiration, systolic blood pressure, diastolic blood pressure and oxygen saturation are recorded.

Progressive Relaxation Exercises: All muscles in the body contract and relax in a coordinated manner. Progressive relaxation exercises, which have been studied in cancer pain, for symptom control in cancer patients receiving chemotherapy, for improving nausea and vomiting after chemotherapy, and for improving quality of life, have been adopted to reduce anxiety, pain, and other stress symptoms, and to increase mental health. The exercise involves systematically tensing and relaxing our muscles. In this way, the exact location of the muscles and their state of tension are known.

Collection of Data:

The data will be obtained from postpartum women who gave birth by cesarean section in the gynecology service of Şanlıurfa Training and Research Hospital and meet the sample selection criteria. Before the application, an explanation will be given to the postpartum women about the purpose of the research, and if they volunteer, their verbal and written permission will be obtained through the "Informed Volunteer Consent Form". Information about postpartum women will be collected by the researcher.

Application of Research

Experimental Group:

Postpartum women will be informed about the research and their written and verbal permissions will be obtained.

Information about postpartum women will be recorded. Women who gave birth by cesarean section who agree to participate in the study will be assigned to 2 groups by randomization method: experimental (group to which progressive relaxation exercises will be applied) and control (group to which progressive relaxation exercises will not be applied).

Progressive relaxation exercises will be explained and taught to the puerperant after cesarean section. Experimental Group (in the group where progressive relaxation exercises were applied); The first application will be made at the 8th postoperative hour. Before the application, the Puerperal Identification Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled out. Starting from the 8th post-op hour, the second and third application will be made eight hours apart within a 48-hour period. On the second day, progressive relaxation exercises will be performed once, twice and three times at eight-hour intervals. At the end of the second day, the Postpartum Definition Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled in again (posttest).

The patient is placed in a supine position. First, the right palm is placed just below the navel, the left hand is placed on the chest and the eyes are closed.

Before inhaling, the lungs are emptied thoroughly by exhaling. When exhaling, the lungs should not be strained and the breath should come out on its own without being forced.

When you start breathing, the lung capacity is divided into two imaginary and the lung is filled completely by counting "one" and "two". Wait for a short time, count "one-two" and evacuate in twice the time you breathe. The right hand should feel the breastbones opening to the side, like a movable bridge31. Wait two seconds before taking another breath.

Take another deep breath and repeat the same process. After repeating slow and deep breathing exercises a few times, progressive relaxation exercises should be started.

In progressive relaxation exercises, all major muscles, in order from bottom to top; right foot, left foot, right leg, left leg, hip, abdominal muscles, back muscles, chest muscles, right hand, left hand, right arm, left arm, neck, shoulders and facial muscles contract while breathing slowly, then exhale It is released by loosening while giving After each muscle contraction and relaxation process, slow and deep breathing exercises should be performed 4-5 times in between before moving on to a new muscle group.

After the relaxation exercises are done and completed in all muscle groups, all muscles contract simultaneously while inhaling and relaxed simultaneously while exhaling. Then, the progressive relaxation exercise is completed with several deep breathing movements.

Control Group:

No application will be carried out with the participants in the control group. At the 8th postoperative hour, the Puerperal Identification Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled out. These participants will be asked not to engage in regular physical activity or sports for 2 days and not to make any changes in their living habits.

During the interview two days later, the Postpartum Identification Form, Beck Anxiety Scale, Visual Analogue Scale (VAS) and Physiological Parameters forms will be filled out again by the puerperant women.

Evaluation of Data

Evaluation of the data obtained as a result of the research will be analyzed using the SPSS (Statistical Package For Social Sciences) 25.0 package program.

Limitation of the Study: It is limited to women who gave birth by cesarean section at Şanlıurfa Training and Research Hospital affiliated with Şanlıurfa Provincial Health Directorate.

Ethical and Legal Aspects of Research Permission will be obtained from Atatürk University Clinical Research Ethics Committee before data collection. Institutional permission will be obtained from Şanlıurfa Provincial Health Directorate. Before the application, verbal and written consent will be obtained from women who gave birth by cesarean section through the "Informed Volunteer Consent Form", if they volunteer, by explaining the purpose of the research.

ELIGIBILITY:
Inclusion criteria; of postpartum women;

1. Being between the ages of 20-35,
2. Primiparous pregnancy
3. Having a transverse cesarean section,
4. It should be taken at the 8th hour postoperatively: since mobilization occurs at the 6th hour after the surgery, it should be taken from the 8th hour postoperatively to prevent fatigue in the woman's extremities and to avoid any health problems (nausea-vomiting, headache-waistache) that prevent her from doing the exercises.
5. Primary school graduate,
6. No mental disability or communication problems. Exclusion criteria;

1. Those who have an open wound on their body and/or a diagnosis of allergic disease on their skin, 2. Puerperal complications (bleeding, infection, fever), 3. Those with cardiac arrhythmia and a pacemaker, 4. At risk of experiencing convulsions; Those with diseases such as eclampsia and epilepsy, 5. Those with kidney or liver disease, 6. Those who have practiced progressive relaxation exercises before, 7. Morbidly obese (BKI over 40), 8. Women using chronic opioids, antidepressants, and psychoactive drugs were not included in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Beck Anxiety Scale | The first application (pretest) was performed at the eighth hour after surgery and The second application (posttest) will be applied at the end of two days.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | The first application (pretest) was performed at the eighth hour after surgery and The second application (posttest) will be applied at the end of two days.

IPD SHARING:
Plan to Share IPD: No